CLINICAL TRIAL: NCT04752293
Title: Pediatric Hypertension and the Renin-Angiotensin SystEm (PHRASE): The Role of Angiotensin-(1-7) in Hypertension and Hypertension-Induced Heart and Kidney Damage
Brief Title: Pediatric Hypertension and the Renin-Angiotensin SystEm (PHRASE)
Acronym: PHRASE
Status: Recruiting | Type: Observational
Sponsor: Wake Forest University Health Sciences (Other)
Collaborators: National Heart, Lung, and Blood Institute (NHLBI) (NIH)
Responsible Party: Sponsor
Other Study IDs: IRB00068679; 1K23HL148394-01A1 (NIH)
Record Dates: First submitted 2021-01-21; First posted 2021-02-12 (Actual); Last update posted 2025-12-11 (Actual); Status verified 2025-12

CONDITIONS: Hypertension; Left Ventricular Hypertrophy; Left Ventricular Dysfunction; Left Atrial Dilatation; Left Ventricular Diastolic Dysfunction; Kidney Diseases; Kidney Injury; Kidney Dysfunction; Sodium Urine High; Blood Pressure Disorders; Uric Acid Retention; Angiotensin Hypertension; Autonomic Dysfunction; Autonomic Imbalance; Pediatric Kidney Disease; Pediatric Obesity; Proteinuria; Albuminuria
Keywords: High Blood Pressure; Elevated Blood Pressure; Hypertension; Pediatric Hypertension; Target Organ Damage; Left Ventricular Hypertrophy; Albuminuria; Uric Acid; Klotho; Fibroblast Growth Factor 23; Renin-Angiotensin-Aldosterone System; Renin-Angiotensin System; Angiotensin-(1-7); Angiotensin II; Angiotensin-Converting Enzyme 2; Angiotensin-Converting Enzyme; Causal Inference; Causal Mediation Analysis; Sensitivity Analysis; Predictive Analysis; Left Ventricular Diastolic Dysfunction; Kidney Injury; Heart Rate Variability; Sodium; Pediatric Obesity; Lifecourse; Kidney Function; Ambulatory Blood Pressure Monitoring; Echocardiogram
MeSH Terms: conditions — Hypertension; Hypertrophy, Left Ventricular; Ventricular Dysfunction, Left; Kidney Diseases; Hyperuricemia; Primary Dysautonomias; Pediatric Obesity; Proteinuria; Albuminuria

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Collecting blood, urine, and saliva samples from participants in the Hypertension Cohort and the Control Cohort. Banking sub-samples of blood, urine, and saliva for future analysis, including for omics-based research (genomics, proteomics, etc.)
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Hypertension Cohort: Participants with newly diagnosed primary hypertension
- Control Cohort: Healthy participants with normal blood pressure

SUMMARY:
Studying the causal roles of components of the renin-angiotensin-aldosterone system (including angiotensin-(1-7) (Ang-(1-7)), angiotensin-converting enzyme 2 (ACE2), Ang II, and ACE), uric acid, and klotho in pediatric hypertension and related target organ injury, including in the heart, kidneys, vasculature, and brain. Recruiting children with a new hypertension diagnosis over a 2-year period from the Hypertension and Pediatric Nephrology Clinics affiliated with Brenner Children's Hospital at Atrium Health Wake Forest Baptist and Atrium Health Levine Children's Hospital. Healthy control participants will be recruited from local general primary care practices. Collecting blood and urine samples to analyze components of the renin-angiotensin-aldosterone system (Ang-(1-7), ACE2, Ang II, ACE), uric acid, and klotho, and measuring blood pressure, heart structure and function, autonomic function, vascular function, and kidney function at baseline, year 1, and year 2. Objectives are to investigate phenotypic and treatment response variability and to causally infer if Ang-(1-7), ACE2, Ang II, ACE, uric acid, and klotho contribute to target organ injury due to hypertension.

DETAILED DESCRIPTION:
This longitudinal prospective cohort study is recruiting children and adolescents aged 7-18 years with newly diagnosed primary hypertension over a 2-year period from the Hypertension and Pediatric Nephrology Clinics affiliated with Brenner Children's Hospital at Atrium Health Wake Forest Baptist, which sees over 300 new patients a year, and the Pediatric Nephrology Clinic at Atrium Health Levine Children's Hospital (Hypertension Cohort). Also recruiting healthy control participants aged 7-18 years with normal blood pressure from local primary care practices (Control Cohort). Collecting blood and urine to analyze Ang-(1-7), ACE2, Ang II, ACE, uric acid, and klotho and measuring pediatric-specific outcomes (blood pressure (casual and ambulatory monitoring), indices of heart structure and function on echocardiogram (left ventricular systolic and diastolic function, left ventricular hypertrophy, etc.), kidney function (creatinine, estimated glomerular filtration rate, albuminuria, proteinuria, urine sodium/potassium), autonomic function (heart rate variability, blood pressure variability, baroreflex sensitivity), and vascular function (arterial stiffness, augmentation index)) at baseline and year 1 (Hypertension Cohort and Control Cohort) and year 2 (Hypertension Cohort). The objectives are to investigate if Ang-(1-7), ACE2, Ang II, and ACE identify phenotypic and treatment response variability and to causally infer if Ang-(1-7), ACE2, Ang II, ACE, uric acid, and klotho contribute to target organ injury, with these Specific Aims:

Aim 1:

(1) Determine if plasma Ang-(1-7) or urine Ang-(1-7)/creatinine differ between the Hypertension vs. Control Cohorts and (2) assess if plasma Ang-(1-7) or urine Ang-(1-7)/creatinine mediate the effect of lisinopril-induced blood pressure reduction on the outcomes (change in heart function and structure, autonomic function, vascular function, and kidney function).

Hypothesis 1a: Baseline Ang-(1-7) is lower in the Hypertension vs. Control Cohort.

Hypothesis 1b: Increased Ang-(1-7) levels over time mediate the effect of lisinopril-induced decreased blood pressure on improved outcomes over 2 years in the Hypertension Cohort.

Aim 2:

(1) Evaluate if plasma Ang-(1-7) or urine Ang-(1-7)/creatinine predict treatment response in participants in the Hypertension Cohort (change in casual blood pressure, ambulatory blood pressure, heart function/structure, autonomic function, vascular function, and kidney function); (2) compare to plasma renin activity and aldosterone; and (3) employ sensitivity analyses to quantify the impact of unmeasured confounding.

Hypothesis 2: Lower baseline Ang-(1-7) predicts greater outcome improvements in the Hypertension Cohort with lower unmeasured confounding and with greater predictive ability compared to plasma renin activity and aldosterone.

Aim 3:

Determine if plasma Ang-(1-7) or urine Ang-(1-7)/creatinine mediate the effects of uric acid and klotho on the outcomes in participants in the Hypertension Cohort. (1) Apply causal mediation to estimate if plasma Ang-(1-7) mediates the effects of uric acid on the outcomes (change in casual blood pressure, ambulatory blood pressure, heart function/structure, autonomic function, and vascular function). (2) Apply causal mediation to estimate if urine Ang-(1-7)/creatinine mediates the effects of klotho on the outcomes (change in casual blood pressure, ambulatory blood pressure, and kidney function).

Hypothesis 3a: Lower plasma Ang-(1-7) mediates the effect of high uric acid on the outcomes in the Hypertension Cohort.

Hypothesis 3b: Lower urine Ang-(1-7)/creatinine mediates the effect of low klotho on the outcomes in the Hypertension Cohort.

Anticipated results have great potential to impact patient care by establishing Ang-(1-7), ACE2, Ang II, and ACE as biomarkers of treatment response, by establishing how Ang-(1-7) and other components of the renin-angiotensin-aldosterone system change in response to an ACE inhibitor, by indicating which patients would benefit most from ACE inhibitors, by identifying novel etiologies of hypertension centered on alterations to the renin-angiotensin-aldosterone system, uric acid, and klotho, and by leading to novel treatments. Indeed, these have been questions of great interest during the COVID-19 pandemic, as ACE2 is the binding site for Severe acute respiratory syndrome (SARS)-CoV-2. Ultimately, the results from this study will improve patient outcomes by promoting cardiovascular health and preventing cardiovascular disease across the lifecourse.

ELIGIBILITY:
INCLUSION CRITERIA: HYPERTENSION COHORT

* 7-18 years of age at time of enrollment
* Confirmed new diagnosis of primary hypertension: no identifiable secondary cause, referred to hypertension or nephrology clinic

  * Age <13 years: BP ≥95th %ile or ≥130/80 mmHg (whichever is lower)
  * Age ≥13 years: BP ≥130/80 mmHg
* Participants and their caregivers must be willing and able to commit to completing the study assessments

EXCLUSION CRITERIA: HYPERTENSION COHORT

* <7 years or >18 years of age at time of enrollment
* BP confirmed as normal or in the elevated BP category based on ≥3 prior office BP measurements on separate days;

  * Age <13 years: BP <95th %ile or <130/80 mmHg (whichever is lower)
  * Age ≥13 years: BP <130/80 mmHg
* A confirmed secondary cause of hypertension
* Confounding medical condition (heart or kidney disease [except hypertension-associated heart changes on echocardiogram or albuminuria], vascular/inflammatory disease, or diabetes)
* Inability to complete study assessments
* Non-English/Spanish speakers
* Current pregnancy
* Ward of the State

INCLUSION CRITERIA: CONTROL COHORT

* 7-18 years of age at time of enrollment
* Normal BP based on ≥3 prior office BP measurements on separate days;

  * Age <13 years: BP <90th %ile or <120/80 mmHg (whichever is lower)
  * Age ≥13 years: BP <120/80 mmHg
* Participants and their caregivers must be willing and able to commit to completing the study assessments

EXCLUSION CRITERIA: CONTROL COHORT

* <7 or >18 years of age at time of enrollment
* Elevated BP or hypertension, based on ≥3 prior office BP measurements on separate days:

  * Age <13 years: BP ≥90th %ile or ≥120/80 mmHg (whichever is lower)
  * Age ≥13 years: BP ≥120/80 mmHg
* History of elevated BP or hypertension
* Current use of BP-lowering medications
* Confounding medical condition (heart or kidney disease, vascular/inflammatory disease, or diabetes)
* Inability to complete study assessments
* Non-English/Spanish speakers
* Current pregnancy
* Ward of the State

Ages: 7 Years to 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Study Population: Hypertension Cohort: Participants will be recruited from among new patients referred to the Hypertension Clinic at Brenner Children's Hospital. Patient population at this clinic, which sees over 300 new patients/year, is 55% White, 25% Black, 16% Hispanic, and 62% male. Goal is to enroll 100 participants over a 2-year period.
  Control Cohort: Participants for this cohort will be recruited from among healthy patients seen at local pediatrics practices. Goal is to enroll 25 participants over a 2-year period, frequency-matched to the Hypertension Cohort on age, self-identified race, and sex.
Sampling Method: Non-Probability Sample
Enrollment: 125 (Estimated)
Dates: Start 2021-05-19 (Actual); Primary Completion 2026-12 (Estimated); Study Completion 2026-12 (Estimated)

PRIMARY OUTCOMES:
Baseline Urine Angiotensin-(1-7)/Creatinine Ratio | Baseline
  Urine angiotensin-(1-7) quantified by a highly developed radioimmunoassay well validated against mass spectrometry and standardized to urine creatinine, quantified by a modified Jaffe assay traceable to isotope dilution mass spectrometry. Report measures of central tendency (e.g., mean, median) and dispersion (e.g., standard deviation, interquartile range, 95 percent confidence interval).
Change in Urine Angiotensin-(1-7)/Creatinine Ratio | Baseline through 2 years
  Urine angiotensin-(1-7) quantified by a highly developed radioimmunoassay well validated against mass spectrometry and standardized to urine creatinine, quantified by a modified Jaffe assay traceable to isotope dilution mass spectrometry. Report measures of central tendency (e.g., mean, median) and dispersion (e.g., standard deviation, interquartile range, 95 percent confidence interval).
Baseline Urine Angiotensin II/Angiotensin-(1-7) Ratio | Baseline
  Urine angiotensin II and angiotensin-(1-7) quantified by highly developed radioimmunoassays well validated against mass spectrometry. Report measures of central tendency (e.g., mean, median) and dispersion (e.g., standard deviation, interquartile range, 95 percent confidence interval).
Change in Urine Angiotensin II/Angiotensin-(1-7) Ratio | Baseline through 2 years
  Urine angiotensin II and angiotensin-(1-7) quantified by highly developed radioimmunoassays well validated against mass spectrometry. Report measures of central tendency (e.g., mean, median) and dispersion (e.g., standard deviation, interquartile range, 95 percent confidence interval).
Baseline Plasma Angiotensin-(1-7) Level | Baseline
  Plasma angiotensin-(1-7) quantified by a highly developed radioimmunoassay well validated against mass spectrometry. Report measures of central tendency (e.g., mean, median) and dispersion (e.g., standard deviation, interquartile range, 95 percent confidence interval).
Change in Plasma Angiotensin-(1-7) Level | Baseline through 2 years
  Plasma angiotensin-(1-7) quantified by a highly developed radioimmunoassay well validated against mass spectrometry. Report measures of central tendency (e.g., mean, median) and dispersion (e.g., standard deviation, interquartile range, 95 percent confidence interval).
Baseline Plasma Angiotensin II/Angiotensin-(1-7) Ratio | Baseline
  Plasma angiotensin II and angiotensin-(1-7) quantified by highly developed radioimmunoassays well validated against mass spectrometry. Report measures of central tendency (e.g., mean, median) and dispersion (e.g., standard deviation, interquartile range, 95 percent confidence interval).
Change in Plasma Angiotensin II/Angiotensin-(1-7) Ratio | Baseline through 2 years
  Plasma angiotensin II and angiotensin-(1-7) quantified by highly developed radioimmunoassays well validated against mass spectrometry. Report measures of central tendency (e.g., mean, median) and dispersion (e.g., standard deviation, interquartile range, 95 percent confidence interval).
Baseline Serum Uric Acid Level | Baseline
  Serum uric acid quantified by a validated uricase assay. Report as a continuous variable with measures of central tendency (e.g., mean) and dispersion (e.g., standard deviation, 95 percent confidence interval).
Change in Serum Uric Acid Level | Baseline through 2 years
  Serum uric acid quantified by a validated uricase assay. Report as a continuous variable with measures of central tendency (e.g., mean) and dispersion (e.g., standard deviation, 95 percent confidence interval).
Baseline Plasma Klotho Level | Baseline
  Plasma α-klotho quantified by a well-validated ELISA. Report measures of central tendency (e.g., mean, median) and dispersion (e.g., standard deviation, interquartile range, 95 percent confidence interval).
Change in Plasma Klotho Level | Baseline through 2 years
  Plasma α-klotho quantified by a well-validated ELISA. Report measures of central tendency (e.g., mean, median) and dispersion (e.g., standard deviation, interquartile range, 95 percent confidence interval).
Baseline Urine Klotho/Creatinine Ratio | Baseline
  Urine α-klotho quantified by a well-validated ELISA and standardized to urine creatinine, quantified by a modified Jaffe assay traceable to isotope dilution mass spectrometry. Report measures of central tendency (e.g., mean, median) and dispersion (e.g., standard deviation, interquartile range, 95 percent confidence interval).
Change in Urine Klotho/Creatinine Ratio | Baseline through 2 years
  Urine α-klotho quantified by a well-validated ELISA and standardized to urine creatinine, quantified by a modified Jaffe assay traceable to isotope dilution mass spectrometry. Report measures of central tendency (e.g., mean, median) and dispersion (e.g., standard deviation, interquartile range, 95 percent confidence interval).
Baseline Manual Systolic Blood Pressure | Baseline
  Average of 3 manual measurements per national guidelines. Report measures of central tendency (e.g., mean) and dispersion (e.g., standard deviation, 95 percent confidence interval).
Change in Manual Systolic Blood Pressure | Baseline through 2 years
  Average of 3 manual measurements per national guidelines. Report measures of central tendency (e.g., mean) and dispersion (e.g., standard deviation, 95 percent confidence interval).
Baseline Manual Diastolic Blood Pressure | Baseline
  Average of 3 manual measurements per national guidelines. Report measures of central tendency (e.g., mean) and dispersion (e.g., standard deviation, 95 percent confidence interval).
Change in Manual Diastolic Blood Pressure | Baseline through 2 years
  Average of 3 manual measurements per national guidelines. Report measures of central tendency (e.g., mean) and dispersion (e.g., standard deviation, 95 percent confidence interval).
Baseline Manual Systolic Blood Pressure Z-score | Baseline
  Average of 3 manual measurements per national guidelines with calculated z-score referenced to normative values by age, sex, and height. Report measures of central tendency (e.g., mean) and dispersion (e.g., standard deviation, 95 percent confidence interval).
Change in Manual Systolic Blood Pressure Z-score | Baseline through 2 years
  Average of 3 manual measurements per national guidelines with calculated z-score referenced to normative values by age, sex, and height. Report measures of central tendency (e.g., mean) and dispersion (e.g., standard deviation, 95 percent confidence interval).
Baseline Manual Diastolic Blood Pressure Z-score | Baseline
  Average of 3 manual measurements per national guidelines with calculated z-score referenced to normative values by age, sex, and height. Report measures of central tendency (e.g., mean) and dispersion (e.g., standard deviation, 95 percent confidence interval).
Change in Manual Diastolic Blood Pressure Z-score | Baseline through 2 years
  Average of 3 manual measurements per national guidelines with calculated z-score referenced to normative values by age, sex, and height. Report measures of central tendency (e.g., mean) and dispersion (e.g., standard deviation, 95 percent confidence interval).
Baseline Ambulatory Systolic Blood Pressure 24-Hour Mean | Baseline
  Measured via ambulatory blood pressure (BP) monitoring. Average systolic BP over a 24-hour period. Report measures of central tendency (e.g., mean, median) and dispersion (e.g., standard deviation, interquartile range, 95 percent confidence interval).
Change in Ambulatory Systolic Blood Pressure 24-Hour Mean | Baseline through 2 years
  Measured via ambulatory blood pressure (BP) monitoring. Average systolic BP over a 24-hour period. Report measures of central tendency (e.g., mean, median) and dispersion (e.g., standard deviation, interquartile range, 95 percent confidence interval).
Baseline Ambulatory Diastolic Blood Pressure 24-Hour Mean | Baseline
  Measured via ambulatory blood pressure (BP) monitoring. Average diastolic BP over a 24-hour period. Report measures of central tendency (e.g., mean, median) and dispersion (e.g., standard deviation, interquartile range, 95 percent confidence interval).
Change in Ambulatory Diastolic Blood Pressure 24-Hour Mean | Baseline through 2 years
  Measured via ambulatory blood pressure (BP) monitoring. Average diastolic BP over a 24-hour period. Report measures of central tendency (e.g., mean, median) and dispersion (e.g., standard deviation, interquartile range, 95 percent confidence interval).
Baseline Left Ventricular Mass Height Index | Baseline
  Left ventricular mass measured via echocardiogram and indexed to height as g/m^2.7. Report measures of central tendency (e.g., mean, median) and dispersion (e.g., standard deviation, interquartile range, 95 percent confidence interval).
Change in Left Ventricular Mass Height Index | Baseline through 2 years
  Left ventricular mass measured via echocardiogram and indexed to height as g/m^2.7. Report measures of central tendency (e.g., mean, median) and dispersion (e.g., standard deviation, interquartile range, 95 percent confidence interval).
Baseline Left Ventricular Mass Body Surface Area Index | Baseline
  Left ventricular mass measured via echocardiogram and indexed to body surface area (BSA) as g/BSA. Report measures of central tendency (e.g., mean, median) and dispersion (e.g., standard deviation, interquartile range, 95 percent confidence interval).
Change in Left Ventricular Mass Body Surface Area Index | Baseline through 2 years
  Left ventricular mass measured via echocardiogram and indexed to body surface area (BSA) as g/BSA. Report measures of central tendency (e.g., mean, median) and dispersion (e.g., standard deviation, interquartile range, 95 percent confidence interval).
Baseline Left Ventricular Hypertrophy | Baseline
  Measured via echocardiogram. Binary variable defined as left ventricular mass index (LVMI) >51 g/m^2.7 (all participants), >115 g/body surface area (BSA) (males), or >95 g/BSA (females), per national guidelines. Report relative measures (e.g., risk ratio) and measures of dispersion (e.g., 95 percent confidence interval).
Change in Left Ventricular Hypertrophy | Baseline through 2 years
  Measured via echocardiogram. Binary variable defined as left ventricular mass index (LVMI) >51 g/m^2.7 (all participants), >115 g/body surface area (BSA) (males), or >95 g/BSA (females), per national guidelines. Report relative measures (e.g., risk ratio) and measures of dispersion (e.g., 95 percent confidence interval).
Baseline Urine Albumin/Creatinine Ratio | Baseline
  Measured in fasting first-morning urine samples. Albumin analyzed in the Clinical Laboratory and creatinine analyzed via a modified Jaffe assay traceable to isotope dilution mass spectrometry. Report measures of central tendency (e.g., mean, median) and dispersion (e.g., standard deviation, interquartile range, 95 percent confidence interval).
Change in Urine Albumin/Creatinine Ratio | Baseline through 2 years
  Measured in fasting first-morning urine samples. Albumin analyzed in the Clinical Laboratory and creatinine analyzed via a modified Jaffe assay traceable to isotope dilution mass spectrometry. Report measures of central tendency (e.g., mean, median) and dispersion (e.g., standard deviation, interquartile range, 95 percent confidence interval).
Baseline Albuminuria | Baseline
  Measured in fasting first-morning urine samples. Albumin analyzed in the Clinical Laboratory and creatinine analyzed via a modified Jaffe assay traceable to isotope dilution mass spectrometry. Binary variable defined as an albumin/creatinine ratio >30 mg/g. Report relative measures (e.g., risk ratio) and measures of dispersion (e.g., 95 percent confidence interval).
Change in Albuminuria | Baseline through 2 years
  Measured in fasting first-morning urine samples. Albumin analyzed in the Clinical Laboratory and creatinine analyzed via a modified Jaffe assay traceable to isotope dilution mass spectrometry. Binary variable defined as an albumin/creatinine ratio >30 mg/g. Report relative measures (e.g., risk ratio) and measures of dispersion (e.g., 95 percent confidence interval).
Baseline Serum Creatinine Level | Baseline
  Measured in the serum and analyzed via a modified Jaffe assay traceable to isotope dilution mass spectrometry. Report measures of central tendency (e.g., mean, median) and dispersion (e.g., standard deviation, interquartile range, 95 percent confidence interval).
Change in Serum Creatinine Level | Baseline through 2 years
  Measured in the serum and analyzed via a modified Jaffe assay traceable to isotope dilution mass spectrometry. Report measures of central tendency (e.g., mean, median) and dispersion (e.g., standard deviation, interquartile range, 95 percent confidence interval).
Baseline Estimated Glomerular Filtration Rate | Baseline
  Estimated using validated, non-race-based, age-appropriate equations (modified Schwartz equation and height- and age-based full-age-spectrum equations with serum creatinine (analyzed via a modified Jaffe assay traceable to isotope dilution mass spectrometry) and serum cystatin C (analyzed via the Clinical Laboratory). Report measures of central tendency (e.g., mean, median) and dispersion (e.g., standard deviation, interquartile range, 95 percent confidence interval).
Change in Estimated Glomerular Filtration Rate | Baseline through 2 years
  Estimated using validated, non-race-based, age-appropriate equations (modified Schwartz equation and height- and age-based full-age-spectrum equations with serum creatinine (analyzed via a modified Jaffe assay traceable to isotope dilution mass spectrometry) and serum cystatin C (analyzed via the Clinical Laboratory). Report measures of central tendency (e.g., mean, median) and dispersion (e.g., standard deviation, interquartile range, 95 percent confidence interval).
Baseline Urine Sodium Concentration | Baseline
  Measured sodium and creatinine in fasting, first-morning urine samples. Sodium analyzed in the Clinical Laboratory, and creatinine analyzed via a modified Jaffe assay traceable to isotope dilution mass spectrometry. Report measures of central tendency (e.g., mean, median) and dispersion (e.g., standard deviation, interquartile range, 95 percent confidence interval).
Change in Urine Sodium Concentration | Baseline through 2 years
  Measured sodium and creatinine in fasting, first-morning urine samples. Sodium analyzed in the Clinical Laboratory, and creatinine analyzed via a modified Jaffe assay traceable to isotope dilution mass spectrometry. Report measures of central tendency (e.g., mean, median) and dispersion (e.g., standard deviation, interquartile range, 95 percent confidence interval).
Baseline Urine Sodium/Potassium Ratio | Baseline
  Measured sodium and potassium in fasting, first-morning urine samples and analyzed in the Clinical Laboratory. Report measures of central tendency (e.g., mean, median) and dispersion (e.g., standard deviation, interquartile range, 95 percent confidence interval).
Change in Urine Sodium/Potassium Ratio | Baseline through 2 years
  Measured sodium and potassium in fasting, first-morning urine samples and analyzed in the Clinical Laboratory. Report measures of central tendency (e.g., mean, median) and dispersion (e.g., standard deviation, interquartile range, 95 percent confidence interval).
Baseline Plasma Renin Activity | Baseline
  Measured in the plasma with a well-validated assay. Report measures of central tendency (e.g., mean, median) and dispersion (e.g., standard deviation, interquartile range, 95 percent confidence interval).
Change in Plasma Renin Activity | Baseline through 2 years
  Measured in the plasma with a well-validated assay. Report measures of central tendency (e.g., mean, median) and dispersion (e.g., standard deviation, interquartile range, 95 percent confidence interval).
Baseline Serum Aldosterone Level | Baseline
  Measured in the serum with a well-validated assay. Report measures of central tendency (e.g., mean, median) and dispersion (e.g., standard deviation, interquartile range, 95 percent confidence interval).
Change in Serum Aldosterone Level | Baseline through 2 years
  Measured in the serum with a well-validated assay. Report measures of central tendency (e.g., mean, median) and dispersion (e.g., standard deviation, interquartile range, 95 percent confidence interval).

SECONDARY OUTCOMES:
Baseline Urine Angiotensin II/Creatinine Ratio | Baseline
  Urine angiotensin II quantified by a highly developed radioimmunoassay well validated against mass spectrometry and standardized to urine creatinine, quantified by a modified Jaffe assay traceable to isotope dilution mass spectrometry. Report measures of central tendency (e.g., mean, median) and dispersion (e.g., standard deviation, interquartile range, 95 percent confidence interval).
Change in Urine Angiotensin II/Creatinine Ratio | Baseline through 2 years
  Urine angiotensin II quantified by a highly developed radioimmunoassay well validated against mass spectrometry and standardized to urine creatinine, quantified by a modified Jaffe assay traceable to isotope dilution mass spectrometry. Report measures of central tendency (e.g., mean, median) and dispersion (e.g., standard deviation, interquartile range, 95 percent confidence interval).
Baseline Urine Angiotensin-Converting Enzyme 2 Level | Baseline
  Measure angiotensin-converting enzyme 2 content and enzymatic activity in first-morning urine samples using established fluorescence-based methods. Standardized to urine creatinine, quantified by a modified Jaffe assay traceable to isotope dilution mass spectrometry. Report measures of central tendency (e.g., mean, median) and dispersion (e.g., standard deviation, interquartile range, 95 percent confidence interval).
Change in Urine Angiotensin-Converting Enzyme 2 Level | Baseline through 2 years
  Measure angiotensin-converting enzyme 2 content and enzymatic activity in first-morning urine samples using established fluorescence-based methods. Standardized to urine creatinine, quantified by a modified Jaffe assay traceable to isotope dilution mass spectrometry. Report measures of central tendency (e.g., mean, median) and dispersion (e.g., standard deviation, interquartile range, 95 percent confidence interval).
Baseline Urine Angiotensin-Converting Enzyme Level | Baseline
  Measure angiotensin-converting enzyme content and enzymatic activity in first-morning urine samples using established fluorescence-based methods. Standardized to urine creatinine, quantified by a modified Jaffe assay traceable to isotope dilution mass spectrometry. Report measures of central tendency (e.g., mean, median) and dispersion (e.g., standard deviation, interquartile range, 95 percent confidence interval).
Change in Urine Angiotensin-Converting Enzyme Level | Baseline through 2 years
  Measure angiotensin-converting enzyme content and enzymatic activity in first-morning urine samples using established fluorescence-based methods. Standardized to urine creatinine, quantified by a modified Jaffe assay traceable to isotope dilution mass spectrometry. Report measures of central tendency (e.g., mean, median) and dispersion (e.g., standard deviation, interquartile range, 95 percent confidence interval).
Baseline Urine Angiotensin-Converting Enzyme/Angiotensin-Converting Enzyme 2 Ratio | Baseline
  Measure angiotensin-converting enzyme and angiotensin-converting enzyme 2 content and enzymatic activity in first-morning urine samples using established fluorescence-based methods. Report measures of central tendency (e.g., mean, median) and dispersion (e.g., standard deviation, interquartile range, 95 percent confidence interval).
Change in Urine Angiotensin-Converting Enzyme/Angiotensin-Converting Enzyme 2 Ratio | Baseline through 2 years
  Measure angiotensin-converting enzyme and angiotensin-converting enzyme 2 content and enzymatic activity in first-morning urine samples using established fluorescence-based methods. Report measures of central tendency (e.g., mean, median) and dispersion (e.g., standard deviation, interquartile range, 95 percent confidence interval).
Baseline Plasma Angiotensin II Level | Baseline
  Plasma angiotensin II quantified by a highly developed radioimmunoassay well validated against mass spectrometry. Report measures of central tendency (e.g., mean, median) and dispersion (e.g., standard deviation, interquartile range, 95 percent confidence interval).
Change in Plasma Angiotensin II Level | Baseline through 2 years
  Plasma angiotensin II quantified by a highly developed radioimmunoassay well validated against mass spectrometry. Report measures of central tendency (e.g., mean, median) and dispersion (e.g., standard deviation, interquartile range, 95 percent confidence interval).
Baseline Serum Angiotensin-Converting Enzyme 2 Level | Baseline
  Measure angiotensin-converting enzyme 2 content and enzymatic activity in serum samples using established fluorescence-based methods. Report measures of central tendency (e.g., mean, median) and dispersion (e.g., standard deviation, interquartile range, 95 percent confidence interval).
Change in Serum Angiotensin-Converting Enzyme 2 Level | Baseline through 2 years
  Measure angiotensin-converting enzyme 2 content and enzymatic activity in serum samples using established fluorescence-based methods. Report measures of central tendency (e.g., mean, median) and dispersion (e.g., standard deviation, interquartile range, 95 percent confidence interval).
Baseline Serum Angiotensin-Converting Enzyme Level | Baseline
  Measure angiotensin-converting enzyme content and enzymatic activity in serum samples using established fluorescence-based methods. Report measures of central tendency (e.g., mean, median) and dispersion (e.g., standard deviation, interquartile range, 95 percent confidence interval).
Change in Serum Angiotensin-Converting Enzyme Level | Baseline through 2 years
  Measure angiotensin-converting enzyme content and enzymatic activity in serum samples using established fluorescence-based methods. Report measures of central tendency (e.g., mean, median) and dispersion (e.g., standard deviation, interquartile range, 95 percent confidence interval).
Baseline Serum Angiotensin-Converting Enzyme/Angiotensin-Converting Enzyme 2 Ratio | Baseline
  Measure angiotensin-converting enzyme and angiotensin-converting enzyme 2 content and enzymatic activity in serum samples using established fluorescence-based methods. Report measures of central tendency (e.g., mean, median) and dispersion (e.g., standard deviation, interquartile range, 95 percent confidence interval).
Change in Serum Angiotensin-Converting Enzyme/Angiotensin-Converting Enzyme 2 Ratio | Baseline through 2 years
  Measure angiotensin-converting enzyme and angiotensin-converting enzyme 2 content and enzymatic activity in serum samples using established fluorescence-based methods. Report measures of central tendency (e.g., mean, median) and dispersion (e.g., standard deviation, interquartile range, 95 percent confidence interval).
Baseline Hyperuricemia | Baseline
  Serum uric acid quantified by a validated uricase assay. Hyperuricemia defined as ≥8.0 mg/dl, reported with relative measures (e.g., risk ratio) and measures of dispersion (e.g., 95 percent confidence interval).
Change in Hyperuricemia | Baseline through 2 years
  Serum uric acid quantified by a validated uricase assay. Hyperuricemia defined as ≥8.0 mg/dl, reported with relative measures (e.g., risk ratio) and measures of dispersion (e.g., 95 percent confidence interval).
Baseline Manual Blood Pressure Classification | Baseline
  Based on average of 3 manual blood pressure (BP) measurements per age-specific national guidelines and age, sex, and height-based BP percentile. Categorized as a 4-level ordinal variable: (1) normal, <90th percentile or <120/80 mmHg; (2) elevated BP, ≥90th to <95th percentile or 120-129/<80 mmHg; (3) stage 1 hypertension, ≥95th to <95th percentile + 12 mmHg or 130-139/80-89 mmHg; (4) stage 2 hypertension, ≥95th percentile + 12 mmHg or ≥140/90 mmHg). Report relative measures (e.g., odds ratio) and measures of dispersion (e.g., 95 percent confidence interval).
Change in Manual Blood Pressure Classification | Baseline through 2 years
  Based on average of 3 manual blood pressure (BP) measurements per age-specific national guidelines and age, sex, and height-based BP percentile. Categorized as a 4-level ordinal variable: (1) normal, <90th percentile or <120/80 mmHg; (2) elevated BP, ≥90th to <95th percentile or 120-129/<80 mmHg; (3) stage 1 hypertension, ≥95th to <95th percentile + 12 mmHg or 130-139/80-89 mmHg; (4) stage 2 hypertension, ≥95th percentile + 12 mmHg or ≥140/90 mmHg). Report relative measures (e.g., odds ratio) and measures of dispersion (e.g., 95 percent confidence interval).
Baseline Ambulatory Systolic Blood Pressure 24-Hour Load | Baseline
  Measured via ambulatory blood pressure (BP) monitoring. Proportion of systolic BP readings over a 24-hour period that are ≥95th percentile for height per national guidelines. Report measures of central tendency (e.g., mean, median) and dispersion (e.g., standard deviation, interquartile range, 95 percent confidence interval).
Change in Ambulatory Systolic Blood Pressure 24-Hour Load | Baseline through 2 years
  Measured via ambulatory blood pressure (BP) monitoring. Proportion of systolic BP readings over a 24-hour period that are ≥95th percentile for height per national guidelines. Report measures of central tendency (e.g., mean, median) and dispersion (e.g., standard deviation, interquartile range, 95 percent confidence interval).
Baseline Ambulatory Diastolic Blood Pressure 24-Hour Load | Baseline
  Measured via ambulatory blood pressure (BP) monitoring. Proportion of diastolic BP readings over a 24-hour period that are ≥95th percentile for height per national guidelines. Report measures of central tendency (e.g., mean, median) and dispersion (e.g., standard deviation, interquartile range, 95 percent confidence interval).
Change in Ambulatory Diastolic Blood Pressure 24-Hour Load | Baseline through 2 years
  Measured via ambulatory blood pressure (BP) monitoring. Proportion of diastolic BP readings over a 24-hour period that are ≥95th percentile for height per national guidelines. Report measures of central tendency (e.g., mean, median) and dispersion (e.g., standard deviation, interquartile range, 95 percent confidence interval).
Baseline Ambulatory Systolic Blood Pressure 24-Hour Index | Baseline
  Measured via ambulatory blood pressure (BP) monitoring. Defined as mean BP over 24-hour period divided by the 95th percentile for sex and height, per national guidelines. Report measures of central tendency (e.g., mean, median) and dispersion (e.g., standard deviation, interquartile range, 95 percent confidence interval).
Change in Ambulatory Systolic Blood Pressure 24-Hour Index | Baseline through 2 years
  Measured via ambulatory blood pressure (BP) monitoring. Defined as mean BP over 24-hour period divided by the 95th percentile for sex and height, per national guidelines. Report measures of central tendency (e.g., mean, median) and dispersion (e.g., standard deviation, interquartile range, 95 percent confidence interval).
Baseline Ambulatory Diastolic Blood Pressure 24-Hour Index | Baseline
  Measured via ambulatory blood pressure (BP) monitoring. Defined as mean BP over 24-hour period divided by the 95th percentile for sex and height, per national guidelines. Report measures of central tendency (e.g., mean, median) and dispersion (e.g., standard deviation, interquartile range, 95 percent confidence interval).
Change in Ambulatory Diastolic Blood Pressure 24-Hour Index | Baseline through 2 years
  Measured via ambulatory blood pressure (BP) monitoring. Defined as mean BP over 24-hour period divided by the 95th percentile for sex and height, per national guidelines. Report measures of central tendency (e.g., mean, median) and dispersion (e.g., standard deviation, interquartile range, 95 percent confidence interval).
Baseline Ambulatory Systolic Blood Pressure Awake Mean | Baseline
  Measured via ambulatory blood pressure (BP) monitoring. Average systolic BP while awake. Report measures of central tendency (e.g., mean, median) and dispersion (e.g., standard deviation, interquartile range, 95 percent confidence interval).
Change in Ambulatory Systolic Blood Pressure Awake Mean | Baseline through 2 years
  Measured via ambulatory blood pressure (BP) monitoring. Average systolic BP while awake. Report measures of central tendency (e.g., mean, median) and dispersion (e.g., standard deviation, interquartile range, 95 percent confidence interval).
Baseline Ambulatory Diastolic Blood Pressure Awake Mean | Baseline
  Measured via ambulatory blood pressure (BP) monitoring. Average diastolic BP while awake. Report measures of central tendency (e.g., mean, median) and dispersion (e.g., standard deviation, interquartile range, 95 percent confidence interval).
Change in Ambulatory Diastolic Blood Pressure Awake Mean | Baseline through 2 years
  Measured via ambulatory blood pressure (BP) monitoring. Average diastolic BP while awake. Report measures of central tendency (e.g., mean, median) and dispersion (e.g., standard deviation, interquartile range, 95 percent confidence interval).
Baseline Ambulatory Systolic Blood Pressure Awake Load | Baseline
  Measured via ambulatory blood pressure (BP) monitoring. Proportion of systolic BP readings while awake that are ≥95th percentile for height per national guidelines. Report measures of central tendency (e.g., mean, median) and dispersion (e.g., standard deviation, interquartile range, 95 percent confidence interval).
Change in Ambulatory Systolic Blood Pressure Awake Load | Baseline through 2 years
  Measured via ambulatory blood pressure (BP) monitoring. Proportion of systolic BP readings while awake that are ≥95th percentile for height per national guidelines. Report measures of central tendency (e.g., mean, median) and dispersion (e.g., standard deviation, interquartile range, 95 percent confidence interval).
Baseline Ambulatory Diastolic Blood Pressure Awake Load | Baseline
  Measured via ambulatory blood pressure (BP) monitoring. Proportion of diastolic BP readings while awake that are ≥95th percentile for height per national guidelines. Report measures of central tendency (e.g., mean, median) and dispersion (e.g., standard deviation, interquartile range, 95 percent confidence interval).
Change in Ambulatory Diastolic Blood Pressure Awake Load | Baseline through 2 years
  Measured via ambulatory blood pressure (BP) monitoring. Proportion of diastolic BP readings while awake that are ≥95th percentile for height per national guidelines. Report measures of central tendency (e.g., mean, median) and dispersion (e.g., standard deviation, interquartile range, 95 percent confidence interval).
Baseline Ambulatory Systolic Blood Pressure Awake Index | Baseline
  Measured via ambulatory blood pressure (BP) monitoring. Defined as mean BP while awake divided by the 95th percentile for sex and height, per national guidelines. Report measures of central tendency (e.g., mean, median) and dispersion (e.g., standard deviation, interquartile range, 95 percent confidence interval).
Change in Ambulatory Systolic Blood Pressure Awake Index | Baseline through 2 years
  Measured via ambulatory blood pressure (BP) monitoring. Defined as mean BP while awake divided by the 95th percentile for sex and height, per national guidelines. Report measures of central tendency (e.g., mean, median) and dispersion (e.g., standard deviation, interquartile range, 95 percent confidence interval).
Baseline Ambulatory Diastolic Blood Pressure Awake Index | Baseline
  Measured via ambulatory blood pressure (BP) monitoring. Defined as mean BP while awake divided by the 95th percentile for sex and height, per national guidelines. Report measures of central tendency (e.g., mean, median) and dispersion (e.g., standard deviation, interquartile range, 95 percent confidence interval).
Change in Ambulatory Diastolic Blood Pressure Awake Index | Baseline through 2 years
  Measured via ambulatory blood pressure (BP) monitoring. Defined as mean BP while awake divided by the 95th percentile for sex and height, per national guidelines. Report measures of central tendency (e.g., mean, median) and dispersion (e.g., standard deviation, interquartile range, 95 percent confidence interval).
Baseline Ambulatory Systolic Blood Pressure Asleep Mean | Baseline
  Measured via ambulatory blood pressure (BP) monitoring. Average systolic BP while asleep. Report measures of central tendency (e.g., mean, median) and dispersion (e.g., standard deviation, interquartile range, 95 percent confidence interval).
Change in Ambulatory Systolic Blood Pressure Asleep Mean | Baseline through 2 years
  Measured via ambulatory blood pressure (BP) monitoring. Average systolic BP while asleep. Report measures of central tendency (e.g., mean, median) and dispersion (e.g., standard deviation, interquartile range, 95 percent confidence interval).
Baseline Ambulatory Diastolic Blood Pressure Asleep Mean | Baseline
  Measured via ambulatory blood pressure (BP) monitoring. Average diastolic BP while asleep. Report measures of central tendency (e.g., mean, median) and dispersion (e.g., standard deviation, interquartile range, 95 percent confidence interval).
Change in Ambulatory Diastolic Blood Pressure Asleep Mean | Baseline through 2 years
  Measured via ambulatory blood pressure (BP) monitoring. Average diastolic BP while asleep. Report measures of central tendency (e.g., mean, median) and dispersion (e.g., standard deviation, interquartile range, 95 percent confidence interval).
Baseline Ambulatory Systolic Blood Pressure Asleep Load | Baseline
  Measured via ambulatory blood pressure (BP) monitoring. Proportion of systolic BP readings while asleep that are ≥95th percentile for height per national guidelines. Report measures of central tendency (e.g., mean, median) and dispersion (e.g., standard deviation, interquartile range, 95 percent confidence interval).
Change in Ambulatory Systolic Blood Pressure Asleep Load | Baseline through 2 years
  Measured via ambulatory blood pressure (BP) monitoring. Proportion of systolic BP readings while asleep that are ≥95th percentile for height per national guidelines. Report measures of central tendency (e.g., mean, median) and dispersion (e.g., standard deviation, interquartile range, 95 percent confidence interval).
Baseline Ambulatory Diastolic Blood Pressure Asleep Load | Baseline
  Measured via ambulatory blood pressure (BP) monitoring. Proportion of diastolic BP readings while asleep that are ≥95th percentile for height per national guidelines. Report measures of central tendency (e.g., mean, median) and dispersion (e.g., standard deviation, interquartile range, 95 percent confidence interval).
Change in Ambulatory Diastolic Blood Pressure Asleep Load | Baseline through 2 years
  Measured via ambulatory blood pressure (BP) monitoring. Proportion of diastolic BP readings while asleep that are ≥95th percentile for height per national guidelines. Report measures of central tendency (e.g., mean, median) and dispersion (e.g., standard deviation, interquartile range, 95 percent confidence interval).
Baseline Ambulatory Systolic Blood Pressure Asleep Index | Baseline
  Measured via ambulatory blood pressure (BP) monitoring. Defined as mean BP while asleep divided by the 95th percentile for sex and height, per national guidelines. Report measures of central tendency (e.g., mean, median) and dispersion (e.g., standard deviation, interquartile range, 95 percent confidence interval).
Change in Ambulatory Systolic Blood Pressure Asleep Index | Baseline through 2 years
  Measured via ambulatory blood pressure (BP) monitoring. Defined as mean BP while asleep divided by the 95th percentile for sex and height, per national guidelines. Report measures of central tendency (e.g., mean, median) and dispersion (e.g., standard deviation, interquartile range, 95 percent confidence interval).
Baseline Ambulatory Diastolic Blood Pressure Asleep Index | Baseline
  Measured via ambulatory blood pressure (BP) monitoring. Defined as mean BP while asleep divided by the 95th percentile for sex and height, per national guidelines. Report measures of central tendency (e.g., mean, median) and dispersion (e.g., standard deviation, interquartile range, 95 percent confidence interval).
Change in Ambulatory Diastolic Blood Pressure Asleep Index | Baseline through 2 years
  Measured via ambulatory blood pressure (BP) monitoring. Defined as mean BP while asleep divided by the 95th percentile for sex and height, per national guidelines. Report measures of central tendency (e.g., mean, median) and dispersion (e.g., standard deviation, interquartile range, 95 percent confidence interval).
Baseline Ambulatory Systolic Blood Pressure Nocturnal Dipping | Baseline
  Measured via ambulatory blood pressure (BP) monitoring. Proportion calculated as ([ mean awake - mean asleep systolic BP ] / [mean awake systolic BP ]) x 100, per national guidelines. Report measures of central tendency (e.g., mean, median) and dispersion (e.g., standard deviation, interquartile range, 95 percent confidence interval).
Change in Ambulatory Systolic Blood Pressure Nocturnal Dipping | Baseline through 2 years
  Measured via ambulatory blood pressure (BP) monitoring. Proportion calculated as ([ mean awake - mean asleep systolic BP ] / [mean awake systolic BP ]) x 100, per national guidelines. Report measures of central tendency (e.g., mean, median) and dispersion (e.g., standard deviation, interquartile range, 95 percent confidence interval).
Baseline Ambulatory Diastolic Blood Pressure Nocturnal Dipping | Baseline
  Measured via ambulatory blood pressure (BP) monitoring. Proportion calculated as ([ mean awake - mean asleep diastolic BP ] / [mean awake diastolic BP ]) x 100, per national guidelines. Report measures of central tendency (e.g., mean, median) and dispersion (e.g., standard deviation, interquartile range, 95 percent confidence interval).
Change in Ambulatory Diastolic Blood Pressure Nocturnal Dipping | Baseline through 2 years
  Measured via ambulatory blood pressure (BP) monitoring. Proportion calculated as ([ mean awake - mean asleep diastolic BP ] / [mean awake diastolic BP ]) x 100, per national guidelines. Report measures of central tendency (e.g., mean, median) and dispersion (e.g., standard deviation, interquartile range, 95 percent confidence interval).
Baseline Ambulatory Inadequate Nocturnal Dipping | Baseline
  Measured via ambulatory blood pressure (BP) monitoring. Binary variable defined as the proportion of BP nocturnal dipping <10 percent, per national guidelines. Report relative measures (e.g., risk ratio) and measures of dispersion (e.g., 95 percent confidence interval).
Change in Ambulatory Inadequate Nocturnal Dipping | Baseline through 2 years
  Measured via ambulatory blo od pressure (BP) monitoring. Binary variable defined as the proportion of BP nocturnal dipping <10 percent, per national guidelines. Report relative measures (e.g., risk ratio) and measures of dispersion (e.g., 95 percent confidence interval).
Baseline Ambulatory Hypertension | Baseline
  Measured via ambulatory blood pressure (BP) monitoring. Binary variable defined as mean BP ≥95 percentile for height AND load ≥25 percent for any time period, per national guidelines. Report relative measures (e.g., risk ratio) and measures of dispersion (e.g., 95 percent confidence interval).
Change in Ambulatory Hypertension | Baseline through 2 years
  Measured via ambulatory blood pressure (BP) monitoring. Binary variable defined as mean BP ≥95 percentile for height AND load ≥25 percent for any time period, per national guidelines. Report relative measures (e.g., risk ratio) and measures of dispersion (e.g., 95 percent confidence interval).
Baseline Relative Left Ventricular Wall Thickness | Baseline
  Measured via echocardiogram. Report measures of central tendency (e.g., mean, median) and dispersion (e.g., standard deviation, interquartile range, 95 percent confidence interval).
Change in Relative Left Ventricular Wall Thickness | Baseline through 2 years
  Measured via echocardiogram. Report measures of central tendency (e.g., mean, median) and dispersion (e.g., standard deviation, interquartile range, 95 percent confidence interval).
Baseline Elevated Relative Left Ventricular Wall Thickness | Baseline
  Measured via echocardiogram. Binary variable defined as >0.42, per national guidelines. Report relative measures (e.g., risk ratio) and measures of dispersion (e.g., 95 percent confidence interval).
Change in Elevated Relative Left Ventricular Wall Thickness | Baseline through 2 years
  Measured via echocardiogram. Binary variable defined as >0.42, per national guidelines. Report relative measures (e.g., risk ratio) and measures of dispersion (e.g., 95 percent confidence interval).
Baseline Left Ventricular Geometry Classification | Baseline
  Measured via echocardiogram. 4-level ordinal variable defined as (1) normal (normal left ventricular mass index (LVMI) and normal relative left ventricular wall thickness (RLVWT)); 2) concentric remodeling (normal LVMI and high RLVWT); 3) eccentric hypertrophy (high LVMI and normal RLVWT); 4) concentric hypertrophy (high LVMI and high RLVWT), per national guidelines. Report relative measures (e.g., risk ratio, odds ratio) and measures of dispersion (e.g., 95 percent confidence interval).
Change in Left Ventricular Geometry Classification | Baseline through 2 years
  Measured via echocardiogram. 4-level ordinal variable defined as (1) normal (normal left ventricular mass index (LVMI) and normal relative left ventricular wall thickness (RLVWT)); 2) concentric remodeling (normal LVMI and high RLVWT); 3) eccentric hypertrophy (high LVMI and normal RLVWT); 4) concentric hypertrophy (high LVMI and high RLVWT), per national guidelines. Report relative measures (e.g., risk ratio, odds ratio) and measures of dispersion (e.g., 95 percent confidence interval).
Baseline Left Ventricular Systolic Function | Baseline
  Measured via echocardiogram. Report measures of central tendency (e.g., mean, median) with dispersion (e.g., standard deviation, interquartile range, 95 percent confidence interval).
Change in Left Ventricular Systolic Function | Baseline through 2 years
  Measured via echocardiogram. Report measures of central tendency (e.g., mean, median) with dispersion (e.g., standard deviation, interquartile range, 95 percent confidence interval).
Baseline Left Ventricular Diastolic Function | Baseline
  Measured via echocardiogram. Report measures of central tendency (e.g., mean, median) with dispersion (e.g., standard deviation, interquartile range, 95 percent confidence interval).
Change in Left Ventricular Diastolic Function | Baseline through 2 years
  Measured via echocardiogram. Report measures of central tendency (e.g., mean, median) with dispersion (e.g., standard deviation, interquartile range, 95 percent confidence interval).
Baseline Left Atrial Size | Baseline
  Measured via echocardiogram. Report measures of central tendency (e.g., mean, median) with dispersion (e.g., standard deviation, interquartile range, 95 percent confidence interval).
Change in Left Atrial Size | Baseline through 2 years
  Measured via echocardiogram. Report measures of central tendency (e.g., mean, median) with dispersion (e.g., standard deviation, interquartile range, 95 percent confidence interval).
Baseline Left Atrial Enlargement | Baseline
  Measured via echocardiogram. Binary variable defined ≥29 ml/m^2, per national guidelines. Report relative measures (e.g., risk ratio) with measures of dispersion (e.g., 95 percent confidence interval).
Change in Left Atrial Enlargement | Baseline through 2 years
  Measured via echocardiogram. Binary variable defined ≥29 ml/m^2, per national guidelines. Report relative measures (e.g., risk ratio) with measures of dispersion (e.g., 95 percent confidence interval).
Baseline Urine Protein/Creatinine Ratio | Baseline
  Measured in fasting first-morning urine samples. Protein analyzed in the Clinical Laboratory and creatinine analyzed via a modified Jaffe assay traceable to isotope dilution mass spectrometry. Report measures of central tendency (e.g., mean, median) and dispersion (e.g., standard deviation, interquartile range, 95 percent confidence interval).
Change in Urine Protein/Creatinine Ratio | Baseline through 2 years
  Measured in fasting first-morning urine samples. Protein analyzed in the Clinical Laboratory and creatinine analyzed via a modified Jaffe assay traceable to isotope dilution mass spectrometry. Report measures of central tendency (e.g., mean, median) and dispersion (e.g., standard deviation, interquartile range, 95 percent confidence interval).
Baseline Proteinuria | Baseline
  Measured in fasting first-morning urine samples. Protein analyzed in the Clinical Laboratory and creatinine analyzed via a modified Jaffe assay traceable to isotope dilution mass spectrometry. Binary variable defined as a protein/creatinine ratio >0.2 mg/mg. Report relative measures (e.g., risk ratio) and measures of dispersion (e.g., 95 percent confidence interval).
Change in Proteinuria | Baseline through 2 years
  Measured in fasting first-morning urine samples. Protein analyzed in the Clinical Laboratory and creatinine analyzed via a modified Jaffe assay traceable to isotope dilution mass spectrometry. Binary variable defined as a protein/creatinine ratio >0.2 mg/mg. Report relative measures (e.g., risk ratio) and measures of dispersion (e.g., 95 percent confidence interval).
Baseline Serum Cystatin C Level | Baseline
  Measured in the serum and analyzed via the Clinical Laboratory. Report measures of central tendency (e.g., mean, median) and dispersion (e.g., standard deviation, interquartile range, 95 percent confidence interval).
Change in Serum Cystatin C Level | Baseline through 2 years
  Measured in the serum and analyzed via the Clinical Laboratory. Report measures of central tendency (e.g., mean, median) and dispersion (e.g., standard deviation, interquartile range, 95 percent confidence interval).
Baseline Elevated Urine Sodium Concentration | Baseline
  Measured sodium and creatinine in fasting, first-morning urine samples. Sodium analyzed in the Clinical Laboratory, and creatinine analyzed via a modified Jaffe assay traceable to isotope dilution mass spectrometry. Binary variable defined as urine sodium/creatinine ratio >1 mmol/mg. Report relative measures (e.g., risk ratio) and measures of dispersion (e.g., 95 percent confidence interval).
Change in Elevated Urine Sodium Concentration | Baseline through 2 years
  Measured sodium and creatinine in fasting, first-morning urine samples. Sodium analyzed in the Clinical Laboratory, and creatinine analyzed via a modified Jaffe assay traceable to isotope dilution mass spectrometry. Binary variable defined as urine sodium/creatinine ratio >1 mmol/mg. Report relative measures (e.g., risk ratio) and measures of dispersion (e.g., 95 percent confidence interval).
Baseline Elevated Urine Sodium/Potassium Ratio | Baseline
  Measured sodium and potassium in fasting, first-morning urine samples and analyzed in the Clinical Laboratory. Binary variable defined as urine sodium/potassium ratio >1 mmol/mmol. Report relative measures (e.g., risk ratio) and measures of dispersion (e.g., 95 percent confidence interval).
Change in Elevated Urine Sodium/Potassium Ratio | Baseline through 2 years
  Measured sodium and potassium in fasting, first-morning urine samples and analyzed in the Clinical Laboratory. Binary variable defined as urine sodium/potassium ratio >1 mmol/mmol. Report relative measures (e.g., risk ratio) and measures of dispersion (e.g., 95 percent confidence interval).
Low Estimated Glomerular Filtration Rate | Through study completion up to 2 years
  Estimated using validated, non-race-based, age-appropriate equations (modified Schwartz equation and height- and age-based full-age-spectrum equations with serum creatinine (analyzed via a modified Jaffe assay traceable to isotope dilution mass spectrometry) and serum cystatin C (analyzed via the Clinical Laboratory). Defined as <90 ml/min/1.73 m^2. Report relative measures (e.g., risk ratio) and measures of dispersion (e.g., 95 percent confidence interval).
Baseline Urine Uric Acid/Creatinine Ratio | Baseline
  Measured in fasting first-morning urine samples. Uric acid quantified by well-validated uricase assay and creatinine via modified Jaffe assay traceable to isotope dilution mass spectrometry. Report measures of central tendency (e.g., mean, median) and dispersion (e.g., standard deviation, interquartile range, 95 percentile confidence interval).
Change in Urine Uric Acid/Creatinine Ratio | Baseline through 2 years
  Measured in fasting first-morning urine samples. Uric acid quantified by well-validated uricase assay and creatinine via modified Jaffe assay traceable to isotope dilution mass spectrometry. Report measures of central tendency (e.g., mean, median) and dispersion (e.g., standard deviation, interquartile range, 95 percentile confidence interval).
Baseline Urine Uric Acid Per Glomerular Filtration Rate | Baseline
  Measured in fasting first-morning urine and serum samples. Uric acid quantified by well-validated uricase assay and creatinine via modified Jaffe assay traceable to isotope dilution mass spectrometry. Calculated as [urine uric acid x serum creatinine] / [urine creatinine]. Report measures of central tendency (e.g., mean, median) and dispersion (e.g., standard deviation, interquartile range, 95 percentile confidence interval).
Change in Urine Uric Acid Per Glomerular Filtration Rate | Baseline through 2 years
  Measured in fasting first-morning urine and serum samples. Uric acid quantified by well-validated uricase assay and creatinine via modified Jaffe assay traceable to isotope dilution mass spectrometry. Calculated as [urine uric acid x serum creatinine] / [urine creatinine]. Report measures of central tendency (e.g., mean, median) and dispersion (e.g., standard deviation, interquartile range, 95 percentile confidence interval).
Baseline Fractional Excretion of Urine Uric Acid | Baseline
  Measured in fasting first-morning urine and serum samples. Uric acid quantified by well-validated uricase assay and creatinine via modified Jaffe assay traceable to isotope dilution mass spectrometry. Calculated as [urine uric acid x serum creatinine] / [urine creatinine x serum uric acid]. Report measures of central tendency (e.g., mean, median) and dispersion (e.g., standard deviation, interquartile range, 95 percentile confidence interval).
Change in Fractional Excretion of Urine Uric Acid | Baseline through 2 years
  Measured in fasting first-morning urine and serum samples. Uric acid quantified by well-validated uricase assay and creatinine via modified Jaffe assay traceable to isotope dilution mass spectrometry. Calculated as [urine uric acid x serum creatinine] / [urine creatinine x serum uric acid]. Report measures of central tendency (e.g., mean, median) and dispersion (e.g., standard deviation, interquartile range, 95 percentile confidence interval).
Baseline Serum Fibroblast Growth Factor 23 Level | Baseline
  Quantified in serum using a validated ELISA. Report measures of central tendency (e.g., mean, median) and dispersion (e.g., standard deviation, interquartile range, 95 percentile confidence interval).
Change in Serum Fibroblast Growth Factor 23 Level | Baseline through 2 years
  Quantified in serum using a validated ELISA. Report measures of central tendency (e.g., mean, median) and dispersion (e.g., standard deviation, interquartile range, 95 percentile confidence interval).
Baseline Urine Fibroblast Growth Factor 23 Level | Baseline
  Quantified in first-morning urine using a validated ELISA, standardized to urine creatinine quantified by a modified Jaffe assay traceable to isotope dilution mass spectrometry. Report measures of central tendency (e.g., mean, median) and dispersion (e.g., standard deviation, interquartile range, 95 percentile confidence interval).
Change in Urine Fibroblast Growth Factor 23 Level | Baseline through 2 years
  Quantified in first-morning urine using a validated ELISA, standardized to urine creatinine quantified by a modified Jaffe assay traceable to isotope dilution mass spectrometry. Report measures of central tendency (e.g., mean, median) and dispersion (e.g., standard deviation, interquartile range, 95 percentile confidence interval).
Baseline Obesity | Baseline
  Height and weight measured in triplicate and average value recorded. Body mass index calculated and obesity defined per national guidelines as body mass index ≥95th percentile for age and sex or ≥30.0 kg/m^2. Report relative measures (e.g., risk ratio, odds ratio) with measures of dispersion (e.g., 95 percentile confidence interval).
Baseline Dietary Sodium Intake | Baseline
  Estimated dietary sodium intake from self-administered food frequency questionnaire. Report measures of central tendency (e.g., mean, median) with dispersion (e.g., standard deviation, interquartile range, 95 percentile confidence interval)
Baseline Disordered Eating | Baseline
  5-item SCOFF questionnaire. Positive if participant answers yes to 2 or more of the 5 questions. Report relative measures (e.g., risk ratio) with measures of dispersion (e.g., 95 percentile confidence interval).
Change in Disordered Eating | Baseline through 2 years
  5-item SCOFF questionnaire. Positive if participant answers yes to 2 or more of the 5 questions. Report relative measures (e.g., risk ratio) with measures of dispersion (e.g., 95 percentile confidence interval).
Baseline Financial Stress | Baseline
  Assessed with a validated questionnaire consisting of one question measured on a 5-point ordinal scale: 1) not hard at all; 2) not very hard; 3) somewhat hard; 4) hard; 5) very hard. Positive if participant reports somewhat hard, hard, or very hard. Report relative measures (e.g., risk ratio, odds ratio) with measures of dispersion (e.g., 95 percentile confidence interval).
Change in Financial Stress | Baseline through 2 years
  Assessed with a validated questionnaire consisting of one question measured on a 5-point ordinal scale: 1) not hard at all; 2) not very hard; 3) somewhat hard; 4) hard; 5) very hard. Positive if participant reports somewhat hard, hard, or very hard. Report relative measures (e.g., risk ratio, odds ratio) with measures of dispersion (e.g., 95 percentile confidence interval).
Baseline Food Insecurity | Baseline
  Assessed with a validated questionnaire consisting of two questions both scored on a 3-point ordinal scale: 1) never true; 2) sometimes true; 3) often true. Positive if participant reports somewhat true or often true to either question. Report relative measures (e.g., risk ratio) with measures of dispersion (e.g., 95 percentile confidence interval).
Change in Food Insecurity | Baseline through 2 years
  Assessed with a validated questionnaire consisting of two questions both scored on a 3-point ordinal scale: 1) never true; 2) sometimes true; 3) often true. Positive if participant reports somewhat true or often true to either question. Report relative measures (e.g., risk ratio) with measures of dispersion (e.g., 95 percentile confidence interval).
Baseline Transportation Stress | Baseline
  Assessed with a validated questionnaire consisting of two binary questions. Positive if participant reports yes to either question. Report relative measures (e.g., risk ratio) with measures of dispersion (e.g., 95 percentile confidence interval).
Change in Transportation Stress | Baseline through 2 years
  Assessed with a validated questionnaire consisting of two binary questions. Positive if participant reports yes to either question. Report relative measures (e.g., risk ratio) with measures of dispersion (e.g., 95 percentile confidence interval).

CONTACTS AND LOCATIONS:
Overall Officials: Andrew M South, MD, MS, Principal Investigator — Wake Forest Health Sciences
Locations (1):
- Wake Forest Health Sciences, Winston-Salem, North Carolina, United States

IPD SHARING:
Plan to Share IPD: Yes
Individual participant data that underlie the results reported in this article, after de-identification, will be shared with other researchers.
Supporting Information: Study Protocol, SAP, Analytic Code
Time Frame: Beginning 12 months and ending six years following article publication.
Access Criteria: Data will be shared with investigators whose proposed use of the data has been approved by an independent review committee identified for this purpose and who provide a methodologically sound proposal. Data will be shared for meta-analysis of individual participant data and/or to achieve aims in the approved proposal.

REFERENCES:
- [Background] Benjamin EJ, Virani SS, Callaway CW, Chamberlain AM, Chang AR, Cheng S, Chiuve SE, Cushman M, Delling FN, Deo R, de Ferranti SD, Ferguson JF, Fornage M, Gillespie C, Isasi CR, Jimenez MC, Jordan LC, Judd SE, Lackland D, Lichtman JH, Lisabeth L, Liu S, Longenecker CT, Lutsey PL, Mackey JS, Matchar DB, Matsushita K, Mussolino ME, Nasir K, O'Flaherty M, Palaniappan LP, Pandey A, Pandey DK, Reeves MJ, Ritchey MD, Rodriguez CJ, Roth GA, Rosamond WD, Sampson UKA, Satou GM, Shah SH, Spartano NL, Tirschwell DL, Tsao CW, Voeks JH, Willey JZ, Wilkins JT, Wu JH, Alger HM, Wong SS, Muntner P; American Heart Association Council on Epidemiology and Prevention Statistics Committee and Stroke Statistics Subcommittee. Heart Disease and Stroke Statistics-2018 Update: A Report From the American Heart Association. Circulation. 2018 Mar 20;137(12):e67-e492. doi: 10.1161/CIR.0000000000000558. Epub 2018 Jan 31. No abstract available. PMID 29386200
- [Background] Laslett LJ, Alagona P Jr, Clark BA 3rd, Drozda JP Jr, Saldivar F, Wilson SR, Poe C, Hart M. The worldwide environment of cardiovascular disease: prevalence, diagnosis, therapy, and policy issues: a report from the American College of Cardiology. J Am Coll Cardiol. 2012 Dec 25;60(25 Suppl):S1-49. doi: 10.1016/j.jacc.2012.11.002. PMID 23257320
- [Background] Danaei G, Ding EL, Mozaffarian D, Taylor B, Rehm J, Murray CJ, Ezzati M. The preventable causes of death in the United States: comparative risk assessment of dietary, lifestyle, and metabolic risk factors. PLoS Med. 2009 Apr 28;6(4):e1000058. doi: 10.1371/journal.pmed.1000058. Epub 2009 Apr 28. PMID 19399161
- [Background] Lim SS, Vos T, Flaxman AD, Danaei G, Shibuya K, Adair-Rohani H, Amann M, Anderson HR, Andrews KG, Aryee M, Atkinson C, Bacchus LJ, Bahalim AN, Balakrishnan K, Balmes J, Barker-Collo S, Baxter A, Bell ML, Blore JD, Blyth F, Bonner C, Borges G, Bourne R, Boussinesq M, Brauer M, Brooks P, Bruce NG, Brunekreef B, Bryan-Hancock C, Bucello C, Buchbinder R, Bull F, Burnett RT, Byers TE, Calabria B, Carapetis J, Carnahan E, Chafe Z, Charlson F, Chen H, Chen JS, Cheng AT, Child JC, Cohen A, Colson KE, Cowie BC, Darby S, Darling S, Davis A, Degenhardt L, Dentener F, Des Jarlais DC, Devries K, Dherani M, Ding EL, Dorsey ER, Driscoll T, Edmond K, Ali SE, Engell RE, Erwin PJ, Fahimi S, Falder G, Farzadfar F, Ferrari A, Finucane MM, Flaxman S, Fowkes FG, Freedman G, Freeman MK, Gakidou E, Ghosh S, Giovannucci E, Gmel G, Graham K, Grainger R, Grant B, Gunnell D, Gutierrez HR, Hall W, Hoek HW, Hogan A, Hosgood HD 3rd, Hoy D, Hu H, Hubbell BJ, Hutchings SJ, Ibeanusi SE, Jacklyn GL, Jasrasaria R, Jonas JB, Kan H, Kanis JA, Kassebaum N, Kawakami N, Khang YH, Khatibzadeh S, Khoo JP, Kok C, Laden F, Lalloo R, Lan Q, Lathlean T, Leasher JL, Leigh J, Li Y, Lin JK, Lipshultz SE, London S, Lozano R, Lu Y, Mak J, Malekzadeh R, Mallinger L, Marcenes W, March L, Marks R, Martin R, McGale P, McGrath J, Mehta S, Mensah GA, Merriman TR, Micha R, Michaud C, Mishra V, Mohd Hanafiah K, Mokdad AA, Morawska L, Mozaffarian D, Murphy T, Naghavi M, Neal B, Nelson PK, Nolla JM, Norman R, Olives C, Omer SB, Orchard J, Osborne R, Ostro B, Page A, Pandey KD, Parry CD, Passmore E, Patra J, Pearce N, Pelizzari PM, Petzold M, Phillips MR, Pope D, Pope CA 3rd, Powles J, Rao M, Razavi H, Rehfuess EA, Rehm JT, Ritz B, Rivara FP, Roberts T, Robinson C, Rodriguez-Portales JA, Romieu I, Room R, Rosenfeld LC, Roy A, Rushton L, Salomon JA, Sampson U, Sanchez-Riera L, Sanman E, Sapkota A, Seedat S, Shi P, Shield K, Shivakoti R, Singh GM, Sleet DA, Smith E, Smith KR, Stapelberg NJ, Steenland K, Stockl H, Stovner LJ, Straif K, Straney L, Thurston GD, Tran JH, Van Dingenen R, van Donkelaar A, Veerman JL, Vijayakumar L, Weintraub R, Weissman MM, White RA, Whiteford H, Wiersma ST, Wilkinson JD, Williams HC, Williams W, Wilson N, Woolf AD, Yip P, Zielinski JM, Lopez AD, Murray CJ, Ezzati M, AlMazroa MA, Memish ZA. A comparative risk assessment of burden of disease and injury attributable to 67 risk factors and risk factor clusters in 21 regions, 1990-2010: a systematic analysis for the Global Burden of Disease Study 2010. Lancet. 2012 Dec 15;380(9859):2224-60. doi: 10.1016/S0140-6736(12)61766-8. PMID 23245609
- [Background] Saran R, Li Y, Robinson B, Ayanian J, Balkrishnan R, Bragg-Gresham J, Chen JT, Cope E, Gipson D, He K, Herman W, Heung M, Hirth RA, Jacobsen SS, Kalantar-Zadeh K, Kovesdy CP, Leichtman AB, Lu Y, Molnar MZ, Morgenstern H, Nallamothu B, O'Hare AM, Pisoni R, Plattner B, Port FK, Rao P, Rhee CM, Schaubel DE, Selewski DT, Shahinian V, Sim JJ, Song P, Streja E, Kurella Tamura M, Tentori F, Eggers PW, Agodoa LY, Abbott KC. US Renal Data System 2014 Annual Data Report: Epidemiology of Kidney Disease in the United States. Am J Kidney Dis. 2015 Jul;66(1 Suppl 1):Svii, S1-305. doi: 10.1053/j.ajkd.2015.05.001. No abstract available. PMID 26111994
- [Background] Chen X, Wang Y. Tracking of blood pressure from childhood to adulthood: a systematic review and meta-regression analysis. Circulation. 2008 Jun 24;117(25):3171-80. doi: 10.1161/CIRCULATIONAHA.107.730366. Epub 2008 Jun 16. PMID 18559702
- [Background] Hao G, Wang X, Treiber FA, Harshfield G, Kapuku G, Su S. Blood Pressure Trajectories From Childhood to Young Adulthood Associated With Cardiovascular Risk: Results From the 23-Year Longitudinal Georgia Stress and Heart Study. Hypertension. 2017 Mar;69(3):435-442. doi: 10.1161/HYPERTENSIONAHA.116.08312. Epub 2017 Jan 16. PMID 28093467
- [Background] Flynn JT, Kaelber DC, Baker-Smith CM, et al; SUBCOMMITTEE ON SCREENING AND MANAGEMENT OF HIGH BLOOD PRESSURE IN CHILDREN. Clinical Practice Guideline for Screening and Management of High Blood Pressure in Children and Adolescents. Pediatrics. 2017; 140(3):e20171904. Pediatrics. 2017 Dec;140(6):e20173035. doi: 10.1542/peds.2017-3035. No abstract available. PMID 29192011
- [Background] Din-Dzietham R, Liu Y, Bielo MV, Shamsa F. High blood pressure trends in children and adolescents in national surveys, 1963 to 2002. Circulation. 2007 Sep 25;116(13):1488-96. doi: 10.1161/CIRCULATIONAHA.106.683243. Epub 2007 Sep 10. PMID 17846287
- [Background] Assadi F. Effect of microalbuminuria lowering on regression of left ventricular hypertrophy in children and adolescents with essential hypertension. Pediatr Cardiol. 2007 Jan-Feb;28(1):27-33. doi: 10.1007/s00246-006-1390-4. Epub 2007 Feb 16. PMID 17308944
- [Background] Litwin M, Niemirska A, Sladowska-Kozlowska J, Wierzbicka A, Janas R, Wawer ZT, Wisniewski A, Feber J. Regression of target organ damage in children and adolescents with primary hypertension. Pediatr Nephrol. 2010 Dec;25(12):2489-99. doi: 10.1007/s00467-010-1626-7. Epub 2010 Aug 21. PMID 20730452
- [Background] Seeman T, Dostalek L, Gilik J. Control of hypertension in treated children and its association with target organ damage. Am J Hypertens. 2012 Mar;25(3):389-95. doi: 10.1038/ajh.2011.218. Epub 2011 Nov 17. PMID 22089110
- [Background] Samuel JP, Samuels JA, Brooks LE, Bell CS, Pedroza C, Molony DA, Tyson JE. Comparative effectiveness of antihypertensive treatment for older children with primary hypertension: study protocol for a series of n-of-1 randomized trials. Trials. 2016 Jan 8;17:16. doi: 10.1186/s13063-015-1142-y. PMID 26746195
- [Background] Benjamin DK Jr, Smith PB, Jadhav P, Gobburu JV, Murphy MD, Hasselblad V, Baker-Smith C, Califf RM, Li JS. Pediatric antihypertensive trial failures: analysis of end points and dose range. Hypertension. 2008 Apr;51(4):834-40. doi: 10.1161/HYPERTENSIONAHA.107.108886. Epub 2008 Mar 10. PMID 18332283
- [Background] Feber J, Ahmed M. Hypertension in children: new trends and challenges. Clin Sci (Lond). 2010 May 14;119(4):151-61. doi: 10.1042/CS20090544. PMID 20477751
- [Background] Hall JE, Granger JP, do Carmo JM, da Silva AA, Dubinion J, George E, Hamza S, Speed J, Hall ME. Hypertension: physiology and pathophysiology. Compr Physiol. 2012 Oct;2(4):2393-442. doi: 10.1002/cphy.c110058. PMID 23720252
- [Background] Chappell MC, Marshall AC, Alzayadneh EM, Shaltout HA, Diz DI. Update on the Angiotensin converting enzyme 2-Angiotensin (1-7)-MAS receptor axis: fetal programing, sex differences, and intracellular pathways. Front Endocrinol (Lausanne). 2014 Jan 9;4:201. doi: 10.3389/fendo.2013.00201. PMID 24409169
- [Background] South AM, Shaltout HA, Washburn LK, Hendricks AS, Diz DI, Chappell MC. Fetal programming and the angiotensin-(1-7) axis: a review of the experimental and clinical data. Clin Sci (Lond). 2019 Jan 8;133(1):55-74. doi: 10.1042/CS20171550. Print 2019 Jan 15. PMID 30622158
- [Background] Shatat IF, Flynn JT. Relationships between renin, aldosterone, and 24-hour ambulatory blood pressure in obese adolescents. Pediatr Res. 2011 Apr;69(4):336-40. doi: 10.1203/PDR.0b013e31820bd148. PMID 21178817
- [Background] Garin EH, Araya CE. Treatment of systemic hypertension in children and adolescents. Curr Opin Pediatr. 2009 Oct;21(5):600-4. doi: 10.1097/MOP.0b013e32832ff3a7. PMID 19606039
- [Background] Chappell MC. Biochemical evaluation of the renin-angiotensin system: the good, bad, and absolute? Am J Physiol Heart Circ Physiol. 2016 Jan 15;310(2):H137-52. doi: 10.1152/ajpheart.00618.2015. Epub 2015 Oct 16. PMID 26475588
- [Background] Wolkow PP, Bujak-Gizycka B, Jawien J, Olszanecki R, Madej J, Rutowski J, Korbut R. Exogenous Angiotensin I Metabolism in Aorta Isolated from Streptozotocin Treated Diabetic Rats. J Diabetes Res. 2016;2016:4846819. doi: 10.1155/2016/4846819. Epub 2016 Oct 10. PMID 27803936
- [Background] Pendergrass KD, Gwathmey TM, Michalek RD, Grayson JM, Chappell MC. The angiotensin II-AT1 receptor stimulates reactive oxygen species within the cell nucleus. Biochem Biophys Res Commun. 2009 Jun 26;384(2):149-54. doi: 10.1016/j.bbrc.2009.04.126. Epub 2009 May 3. PMID 19409874
- [Background] Dilauro M, Zimpelmann J, Robertson SJ, Genest D, Burns KD. Effect of ACE2 and angiotensin-(1-7) in a mouse model of early chronic kidney disease. Am J Physiol Renal Physiol. 2010 Jun;298(6):F1523-32. doi: 10.1152/ajprenal.00426.2009. Epub 2010 Mar 31. PMID 20357030
- [Background] Benter IF, Yousif MH, Anim JT, Cojocel C, Diz DI. Angiotensin-(1-7) prevents development of severe hypertension and end-organ damage in spontaneously hypertensive rats treated with L-NAME. Am J Physiol Heart Circ Physiol. 2006 Feb;290(2):H684-91. doi: 10.1152/ajpheart.00632.2005. PMID 16403946
- [Background] ESCAPE Trial Group; Wuhl E, Trivelli A, Picca S, Litwin M, Peco-Antic A, Zurowska A, Testa S, Jankauskiene A, Emre S, Caldas-Afonso A, Anarat A, Niaudet P, Mir S, Bakkaloglu A, Enke B, Montini G, Wingen AM, Sallay P, Jeck N, Berg U, Caliskan S, Wygoda S, Hohbach-Hohenfellner K, Dusek J, Urasinski T, Arbeiter K, Neuhaus T, Gellermann J, Drozdz D, Fischbach M, Moller K, Wigger M, Peruzzi L, Mehls O, Schaefer F. Strict blood-pressure control and progression of renal failure in children. N Engl J Med. 2009 Oct 22;361(17):1639-50. doi: 10.1056/NEJMoa0902066. PMID 19846849
- [Background] Simoes E Silva AC, Diniz JS, Regueira Filho A, Santos RA. The renin angiotensin system in childhood hypertension: selective increase of angiotensin-(1-7) in essential hypertension. J Pediatr. 2004 Jul;145(1):93-8. doi: 10.1016/j.jpeds.2004.03.055. PMID 15238914
- [Background] Ferrario CM, Martell N, Yunis C, Flack JM, Chappell MC, Brosnihan KB, Dean RH, Fernandez A, Novikov SV, Pinillas C, Luque M. Characterization of angiotensin-(1-7) in the urine of normal and essential hypertensive subjects. Am J Hypertens. 1998 Feb;11(2):137-46. doi: 10.1016/s0895-7061(97)00400-7. PMID 9524041
- [Background] South AM, Nixon PA, Chappell MC, Diz DI, Russell GB, Snively BM, Shaltout HA, Rose JC, O'Shea TM, Washburn LK. Antenatal corticosteroids and the renin-angiotensin-aldosterone system in adolescents born preterm. Pediatr Res. 2017 Jan;81(1-1):88-93. doi: 10.1038/pr.2016.179. Epub 2016 Sep 16. PMID 27636897
- [Background] South AM, Nixon PA, Chappell MC, Diz DI, Russell GB, Jensen ET, Shaltout HA, O'Shea TM, Washburn LK. Association between preterm birth and the renin-angiotensin system in adolescence: influence of sex and obesity. J Hypertens. 2018 Oct;36(10):2092-2101. doi: 10.1097/HJH.0000000000001801. PMID 29846325
- [Background] South AM, Pao AC, Grimm PC. Subclinical injury in pediatric renal transplant patients: ACE2 and Ang-(1-7) as novel biomarkers [abstract]. Clin Transl Sci 2014; 7:232-3.
- [Background] South AM, Nixon PA, Chappell MC, et al. Preterm adolescents exhibit higher blood pressure and sodium retention with higher uric acid and differential circulating renin-angiotensin system expression [abstract]. FASEB J 2018; 32:883.6
- [Background] South AM, Nixon PN, Chappell MC, et al. Elevated blood pressure and sodium retention in young adults born preterm may reflect uric acid-related suppression of renal angiotensin-(1-7) [abstract]. Pediatric Academic Societies 2018; E-PAS2018:3150.3
- [Background] Shaltout HA, Rose JC, Chappell MC, Diz DI. Angiotensin-(1-7) deficiency and baroreflex impairment precede the antenatal Betamethasone exposure-induced elevation in blood pressure. Hypertension. 2012 Feb;59(2):453-8. doi: 10.1161/HYPERTENSIONAHA.111.185876. Epub 2012 Jan 3. PMID 22215705
- [Background] Washburn LK, Nixon PA, Russell GB, Snively BM, O'Shea TM. Preterm Birth Is Associated with Higher Uric Acid Levels in Adolescents. J Pediatr. 2015 Jul;167(1):76-80. doi: 10.1016/j.jpeds.2015.03.043. Epub 2015 Apr 11. PMID 25868431
- [Background] Shaltout HA, Nixon PA, Chappell MC, et al. Impaired autonomic function in young adults born preterm with very low birth weight is associated with elevated serum uric acid levels [abstract]. Hypertension 2018; ePub; doi:
- [Background] South AM, Nixon PN, Chappell MC, et al. Urinary α-klotho is associated with higher blood pressure and reduced urinary angiotensin-(1-7) in young adults born preterm [abstract]. Pediatric Academic Societies 2018; E-PAS2018:1502.841
- [Background] South AM, Arguelles L, Finer G, Langman CB. Race, obesity, and the renin-angiotensin-aldosterone system: treatment response in children with primary hypertension. Pediatr Nephrol. 2017 Sep;32(9):1585-1594. doi: 10.1007/s00467-017-3665-9. Epub 2017 Apr 14. PMID 28411317
- [Background] Khosla UM, Zharikov S, Finch JL, Nakagawa T, Roncal C, Mu W, Krotova K, Block ER, Prabhakar S, Johnson RJ. Hyperuricemia induces endothelial dysfunction. Kidney Int. 2005 May;67(5):1739-42. doi: 10.1111/j.1523-1755.2005.00273.x. PMID 15840020
- [Background] Viazzi F, Antolini L, Giussani M, Brambilla P, Galbiati S, Mastriani S, Stella A, Pontremoli R, Valsecchi MG, Genovesi S. Serum uric acid and blood pressure in children at cardiovascular risk. Pediatrics. 2013 Jul;132(1):e93-9. doi: 10.1542/peds.2013-0047. Epub 2013 Jun 17. PMID 23776119
- [Background] Feig DI, Soletsky B, Johnson RJ. Effect of allopurinol on blood pressure of adolescents with newly diagnosed essential hypertension: a randomized trial. JAMA. 2008 Aug 27;300(8):924-32. doi: 10.1001/jama.300.8.924. PMID 18728266
- [Background] Zhang JX, Zhang YP, Wu QN, Chen B. Uric acid induces oxidative stress via an activation of the renin-angiotensin system in 3T3-L1 adipocytes. Endocrine. 2015 Feb;48(1):135-42. doi: 10.1007/s12020-014-0239-5. Epub 2014 Mar 28. PMID 24671741
- [Background] Mule G, Castiglia A, Morreale M, Geraci G, Cusumano C, Guarino L, Altieri D, Panzica M, Vaccaro F, Cottone S. Serum uric acid is not independently associated with plasma renin activity and plasma aldosterone in hypertensive adults. Nutr Metab Cardiovasc Dis. 2017 Apr;27(4):350-359. doi: 10.1016/j.numecd.2016.12.008. Epub 2016 Dec 27. PMID 28274727
- [Background] McMullan CJ, Borgi L, Fisher N, Curhan G, Forman J. Effect of Uric Acid Lowering on Renin-Angiotensin-System Activation and Ambulatory BP: A Randomized Controlled Trial. Clin J Am Soc Nephrol. 2017 May 8;12(5):807-816. doi: 10.2215/CJN.10771016. Epub 2017 Mar 20. PMID 28320765
- [Background] South AM, Shaltout HA, Nixon PA, Diz DI, Jensen ET, O'Shea TM, Chappell MC, Washburn LK. Association of circulating uric acid and angiotensin-(1-7) in relation to higher blood pressure in adolescents and the influence of preterm birth. J Hum Hypertens. 2020 Dec;34(12):818-825. doi: 10.1038/s41371-020-0335-3. Epub 2020 Apr 28. PMID 32346123
- [Background] Su XM, Yang W. Klotho protein lowered in elderly hypertension. Int J Clin Exp Med. 2014 Aug 15;7(8):2347-50. eCollection 2014. PMID 25232434
- [Background] Nagai R, Saito Y, Ohyama Y, Aizawa H, Suga T, Nakamura T, Kurabayashi M, Kuroo M. Endothelial dysfunction in the klotho mouse and downregulation of klotho gene expression in various animal models of vascular and metabolic diseases. Cell Mol Life Sci. 2000 May;57(5):738-46. doi: 10.1007/s000180050038. PMID 10892340
- [Background] Karalliedde J, Maltese G, Hill B, Viberti G, Gnudi L. Effect of renin-angiotensin system blockade on soluble Klotho in patients with type 2 diabetes, systolic hypertension, and albuminuria. Clin J Am Soc Nephrol. 2013 Nov;8(11):1899-905. doi: 10.2215/CJN.02700313. Epub 2013 Aug 8. PMID 23929932
- [Background] Mitani H, Ishizaka N, Aizawa T, Ohno M, Usui S, Suzuki T, Amaki T, Mori I, Nakamura Y, Sato M, Nangaku M, Hirata Y, Nagai R. In vivo klotho gene transfer ameliorates angiotensin II-induced renal damage. Hypertension. 2002 Apr;39(4):838-43. doi: 10.1161/01.hyp.0000013734.33441.ea. PMID 11967236
- [Background] Yoon HE, Ghee JY, Piao S, Song JH, Han DH, Kim S, Ohashi N, Kobori H, Kuro-o M, Yang CW. Angiotensin II blockade upregulates the expression of Klotho, the anti-ageing gene, in an experimental model of chronic cyclosporine nephropathy. Nephrol Dial Transplant. 2011 Mar;26(3):800-13. doi: 10.1093/ndt/gfq537. Epub 2010 Sep 2. PMID 20813770
- [Background] Zhou L, Mo H, Miao J, Zhou D, Tan RJ, Hou FF, Liu Y. Klotho Ameliorates Kidney Injury and Fibrosis and Normalizes Blood Pressure by Targeting the Renin-Angiotensin System. Am J Pathol. 2015 Dec;185(12):3211-23. doi: 10.1016/j.ajpath.2015.08.004. Epub 2015 Oct 24. PMID 26475416
- [Background] South AM, Shaltout HA, Gwathmey TM, Jensen ET, Nixon PA, Diz DI, Chappell MC, Washburn LK. Lower urinary alpha-Klotho is associated with lower angiotensin-(1-7) and higher blood pressure in young adults born preterm with very low birthweight. J Clin Hypertens (Greenwich). 2020 Jun;22(6):1033-1040. doi: 10.1111/jch.13897. Epub 2020 May 31. PMID 32475043
- [Background] ClinicalTrials.gov [Internet]. Bethesda (MD): National Library of Medicine (US). 2017/10/10. Identifier NCT03305562: Pediatric Hypertension Registry (PHREG); 2017/10/16. Available from: https://ClinicalTrials.gov/show/NCT03305562
- [Background] ClinicalTrials.gov [Internet]. Bethesday (MD): National Library of Medicine (US). 2017 Oct 16. Identifier NCT03310684: Pediatric Primary Hypertension and the Renin-Angiotensin System (PHRAS); 2017 Oct 16. Available from: https://ClinicalTrials.gov/show/NCT03310684
- [Background] Lytle LA, Nichaman MZ, Obarzanek E, Glovsky E, Montgomery D, Nicklas T, Zive M, Feldman H. Validation of 24-hour recalls assisted by food records in third-grade children. The CATCH Collaborative Group. J Am Diet Assoc. 1993 Dec;93(12):1431-6. doi: 10.1016/0002-8223(93)92247-u. PMID 8245378
- [Background] Morisky DE, Ang A, Krousel-Wood M, Ward HJ. Predictive validity of a medication adherence measure in an outpatient setting. J Clin Hypertens (Greenwich). 2008 May;10(5):348-54. doi: 10.1111/j.1751-7176.2008.07572.x. PMID 18453793
- [Background] Eakin MN, Brady T, Kandasamy V, Fivush B, Riekert KA. Disparities in antihypertensive medication adherence in adolescents. Pediatr Nephrol. 2013 Aug;28(8):1267-73. doi: 10.1007/s00467-013-2455-2. Epub 2013 Mar 20. PMID 23512259
- [Background] Tang KL, Quan H, Rabi DM. Measuring medication adherence in patients with incident hypertension: a retrospective cohort study. BMC Health Serv Res. 2017 Feb 13;17(1):135. doi: 10.1186/s12913-017-2073-y. PMID 28193217
- [Background] Pruette CS, Coburn SS, Eaton CK, Brady TM, Tuchman S, Mendley S, Fivush BA, Eakin MN, Riekert KA. Does a multimethod approach improve identification of medication nonadherence in adolescents with chronic kidney disease? Pediatr Nephrol. 2019 Jan;34(1):97-105. doi: 10.1007/s00467-018-4044-x. Epub 2018 Aug 16. PMID 30116892
- [Background] Loichinger MH, Towner D, Thompson KS, Ahn HJ, Bryant-Greenwood GD. Systemic and placental alpha-klotho: Effects of preeclampsia in the last trimester of gestation. Placenta. 2016 May;41:53-61. doi: 10.1016/j.placenta.2016.03.004. Epub 2016 Mar 8. PMID 27208408
- [Background] Drew DA, Katz R, Kritchevsky S, Ix J, Shlipak M, Gutierrez OM, Newman A, Hoofnagle A, Fried L, Semba RD, Sarnak M. Association between Soluble Klotho and Change in Kidney Function: The Health Aging and Body Composition Study. J Am Soc Nephrol. 2017 Jun;28(6):1859-1866. doi: 10.1681/ASN.2016080828. Epub 2017 Jan 19. PMID 28104822
- [Background] Rosner B, Cook N, Portman R, Daniels S, Falkner B. Determination of blood pressure percentiles in normal-weight children: some methodological issues. Am J Epidemiol. 2008 Mar 15;167(6):653-66. doi: 10.1093/aje/kwm348. Epub 2008 Jan 29. PMID 18230679
- [Background] Flynn JT, Daniels SR, Hayman LL, Maahs DM, McCrindle BW, Mitsnefes M, Zachariah JP, Urbina EM; American Heart Association Atherosclerosis, Hypertension and Obesity in Youth Committee of the Council on Cardiovascular Disease in the Young. Update: ambulatory blood pressure monitoring in children and adolescents: a scientific statement from the American Heart Association. Hypertension. 2014 May;63(5):1116-35. doi: 10.1161/HYP.0000000000000007. Epub 2014 Mar 3. No abstract available. PMID 24591341
- [Background] Sorof JM, Cardwell G, Franco K, Portman RJ. Ambulatory blood pressure and left ventricular mass index in hypertensive children. Hypertension. 2002 Apr;39(4):903-8. doi: 10.1161/01.hyp.0000013266.40320.3b. PMID 11967247
- [Background] Wuhl E, Witte K, Soergel M, Mehls O, Schaefer F; German Working Group on Pediatric Hypertension. Distribution of 24-h ambulatory blood pressure in children: normalized reference values and role of body dimensions. J Hypertens. 2002 Oct;20(10):1995-2007. doi: 10.1097/00004872-200210000-00019. PMID 12359978
- [Background] Khoury PR, Mitsnefes M, Daniels SR, Kimball TR. Age-specific reference intervals for indexed left ventricular mass in children. J Am Soc Echocardiogr. 2009 Jun;22(6):709-14. doi: 10.1016/j.echo.2009.03.003. Epub 2009 May 7. PMID 19423289
- [Background] Khoury M, Khoury PR, Dolan LM, Kimball TR, Urbina EM. Clinical Implications of the Revised AAP Pediatric Hypertension Guidelines. Pediatrics. 2018 Aug;142(2):e20180245. doi: 10.1542/peds.2018-0245. Epub 2018 Jul 5. PMID 29976572
- [Background] Baker-Smith CM, Flinn SK, Flynn JT, Kaelber DC, Blowey D, Carroll AE, Daniels SR, de Ferranti SD, Dionne JM, Falkner B, Gidding SS, Goodwin C, Leu MG, Powers ME, Rea C, Samuels J, Simasek M, Thaker VV, Urbina EM; SUBCOMMITTEE ON SCREENING AND MANAGEMENT OF HIGH BP IN CHILDREN. Diagnosis, Evaluation, and Management of High Blood Pressure in Children and Adolescents. Pediatrics. 2018 Sep;142(3):e20182096. doi: 10.1542/peds.2018-2096. Epub 2018 Aug 20. PMID 30126937
- [Background] Fortunato JE, Tegeler CL, Gerdes L, Lee SW, Pajewski NM, Franco ME, Cook JF, Shaltout HA, Tegeler CH. Use of an allostatic neurotechnology by adolescents with postural orthostatic tachycardia syndrome (POTS) is associated with improvements in heart rate variability and changes in temporal lobe electrical activity. Exp Brain Res. 2016 Mar;234(3):791-8. doi: 10.1007/s00221-015-4499-y. Epub 2015 Dec 8. PMID 26645307
- [Background] Parati G, Saul JP, Di Rienzo M, Mancia G. Spectral analysis of blood pressure and heart rate variability in evaluating cardiovascular regulation. A critical appraisal. Hypertension. 1995 Jun;25(6):1276-86. doi: 10.1161/01.hyp.25.6.1276. PMID 7768574
- [Background] Butlin M, Qasem A. Large Artery Stiffness Assessment Using SphygmoCor Technology. Pulse (Basel). 2017 Jan;4(4):180-192. doi: 10.1159/000452448. Epub 2016 Dec 1. PMID 28229053
- [Background] Rademacher ER, Sinaiko AR. Albuminuria in children. Curr Opin Nephrol Hypertens. 2009 May;18(3):246-51. doi: 10.1097/MNH.0b013e3283294b98. PMID 19276802
- [Background] Schwartz GJ, Schneider MF, Maier PS, Moxey-Mims M, Dharnidharka VR, Warady BA, Furth SL, Munoz A. Improved equations estimating GFR in children with chronic kidney disease using an immunonephelometric determination of cystatin C. Kidney Int. 2012 Aug;82(4):445-53. doi: 10.1038/ki.2012.169. PMID 22622496
- [Background] Schwartz GJ, Munoz A, Schneider MF, Mak RH, Kaskel F, Warady BA, Furth SL. New equations to estimate GFR in children with CKD. J Am Soc Nephrol. 2009 Mar;20(3):629-37. doi: 10.1681/ASN.2008030287. Epub 2009 Jan 21. PMID 19158356
- [Background] Pottel H, Bjork J, Bokenkamp A, Berg U, Asling-Monemi K, Selistre L, Dubourg L, Hansson M, Littmann K, Jones I, Sjostrom P, Nyman U, Delanaye P. Estimating glomerular filtration rate at the transition from pediatric to adult care. Kidney Int. 2019 May;95(5):1234-1243. doi: 10.1016/j.kint.2018.12.020. Epub 2019 Feb 28. PMID 30922665
- [Background] Kuczmarski RJ, Ogden CL, Guo SS, Grummer-Strawn LM, Flegal KM, Mei Z, Wei R, Curtin LR, Roche AF, Johnson CL. 2000 CDC Growth Charts for the United States: methods and development. Vital Health Stat 11. 2002 May;(246):1-190. PMID 12043359
- [Background] Croghan C, Egeghy PP. Methods of dealing with values below the limit of detection using SAS. Southeastern SAS User Group. 2003;N/A
- [Background] Shrier I, Platt RW. Reducing bias through directed acyclic graphs. BMC Med Res Methodol. 2008 Oct 30;8:70. doi: 10.1186/1471-2288-8-70. PMID 18973665
- [Background] Knol MJ, VanderWeele TJ. Recommendations for presenting analyses of effect modification and interaction. Int J Epidemiol. 2012 Apr;41(2):514-20. doi: 10.1093/ije/dyr218. Epub 2012 Jan 9. PMID 22253321
- [Background] Hansen BB, Klopfer SO. Optimal full matching and related designs via network flows. J Comput Graph Stat 2006; 15:609-27.
- [Background] Hansen BB, Fredrickson M, Buckner J, et al. Using Optmatch on data in SAS, Stata, etc. 2019;2019
- [Background] Zhang Z, Zheng C, Kim C, Van Poucke S, Lin S, Lan P. Causal mediation analysis in the context of clinical research. Ann Transl Med. 2016 Nov;4(21):425. doi: 10.21037/atm.2016.11.11. PMID 27942516
- [Background] Lin S-H. 2016. Causal mediation analysis with time-varying and multiple mediators. Doctoral Dissertation, Harvard T.H. Chan School of Public Health.
- [Background] VanderWeele TJ. A unification of mediation and interaction: a 4-way decomposition. Epidemiology. 2014 Sep;25(5):749-61. doi: 10.1097/EDE.0000000000000121. PMID 25000145
- [Background] Washburn LK, Nixon PA, Snively BM, et al. Increased blood pressure and the circulating renin-angiotensin system in adolescents born preterm [abstract]. Pediatric Academic Societies. 2013; ePub; doi:
- [Background] Kim YM, Cologne JB, Cullings HM. Simple power analysis in causal mediation models for a dichotomous outcome based on the mediation proportion. J Korean Data Inf Sci Soc 2017; 28:669-84
- [Background] Jimenez A, Chen A, Lin JJ, South AM. Does MEST-C score predict outcomes in pediatric Henoch-Schonlein purpura nephritis? Pediatr Nephrol. 2019 Dec;34(12):2583-2589. doi: 10.1007/s00467-019-04327-2. Epub 2019 Aug 11. PMID 31402405
- [Background] Pun BT, Balas MC, Barnes-Daly MA, Thompson JL, Aldrich JM, Barr J, Byrum D, Carson SS, Devlin JW, Engel HJ, Esbrook CL, Hargett KD, Harmon L, Hielsberg C, Jackson JC, Kelly TL, Kumar V, Millner L, Morse A, Perme CS, Posa PJ, Puntillo KA, Schweickert WD, Stollings JL, Tan A, D'Agostino McGowan L, Ely EW. Caring for Critically Ill Patients with the ABCDEF Bundle: Results of the ICU Liberation Collaborative in Over 15,000 Adults. Crit Care Med. 2019 Jan;47(1):3-14. doi: 10.1097/CCM.0000000000003482. PMID 30339549
- [Background] Lin DY, Psaty BM, Kronmal RA. Assessing the sensitivity of regression results to unmeasured confounders in observational studies. Biometrics. 1998 Sep;54(3):948-63. PMID 9750244
- [Background] VanderWeele TJ, Ding P. Sensitivity Analysis in Observational Research: Introducing the E-Value. Ann Intern Med. 2017 Aug 15;167(4):268-274. doi: 10.7326/M16-2607. Epub 2017 Jul 11. PMID 28693043
- [Background] Shatat IF, Abdallah RT, Sas DJ, Hailpern SM. Serum uric acid in U.S. adolescents: distribution and relationship to demographic characteristics and cardiovascular risk factors. Pediatr Res. 2012 Jul;72(1):95-100. doi: 10.1038/pr.2012.47. PMID 22465909
- [Background] Writing Group for the Division of Cardiovascular Sciences' Strategic Vision Implementation Plan; Goff DC Jr, Buxton DB, Pearson GD, Wei GS, Gosselin TE, Addou EA, Stoney CM, Desvigne-Nickens P, Srinivas PR, Galis ZS, Pratt C, Kit KBK, Maric-Bilkan C, Nicastro HL, Wong RP, Sachdev V, Chen J, Fine L. Implementing the National Heart, Lung, and Blood Institute's Strategic Vision in the Division of Cardiovascular Sciences. Circ Res. 2019 Feb 15;124(4):491-497. doi: 10.1161/CIRCRESAHA.118.314338. PMID 31031412